CLINICAL TRIAL: NCT05390398
Title: Study on Fatigue in Colorectal Cancer Survivors, a Lifestyle Intervention
Acronym: SoFiT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: World Cancer Research Fund International (Other); Gelderse Vallei Hospital (Other); Flevoziekenhuis (Other); Slingeland Hospital (Other); Rijnstate Hospital (Other); Het Prospectief Landelijk CRC cohort (PLCRC) (Unknown); Deventer Ziekenhuis (Other)
Responsible Party: Principal Investigator, Renate Winkels, Dr.Ir., Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL75999.091.21
Record Dates: First submitted 2022-03-24; First posted 2022-05-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Cancer-related Fatigue; Colon Cancer; Rectal Cancer
Keywords: Intervention study; Randomized controlled trial; Lifestyle; Behaviour change; Colorectal cancer survivors; Cancer-related fatigue; Lifestyle coach; Nutrition; Physical activity; Skeletal muscle fat infiltration
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two parallel arms: intervention and control.
Who Masked: Outcomes Assessor
Masking Description: The nature of the intervention does not allow for blinding of the participants or researchers. The baseline measurements are however blinded as both the participant and the researchers do not yet know in which group the participant will be classified. Randomization is done directly after the baseline measurements. After data collection, the database will be coded by an independent researcher to ensure that data analysis is conducted in a blinded way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group follows a six-month personalized lifestyle program to increase adherence to the World Cancer Research Fund cancer prevention guidelines on healthy nutrition, physical activity and healthy weight.
  Interventions: Behavioral: Behaviour change guided lifestyle intervention
- Wait-list usual care group (No Intervention): The wait-list usual care group follows usual care and usual activities. Participants receive a lifestyle program after the intervention period of six months: this includes two personalized behavioural coaching sessions and any material that the intervention group also received.

INTERVENTIONS:
Behavioral: Behaviour change guided lifestyle intervention — Participants in the intervention group receive personalized coaching from a lifestyle coach on adhering to the World Cancer Research Fund cancer prevention guidelines. The lifestyle coach is specialized in behaviour change techniques and uses these as the core of the lifestyle coaching. For each participant behavioural determinants will be assessed and targeted with specific applicable behaviour change techniques.
  Arms: Intervention group

SUMMARY:
The SoFiT study is a randomized controlled trial examining the effects of a behaviour change guided lifestyle intervention on increasing adherence to the World Cancer Research Fund cancer prevention guidelines, compared to the wait-list usual care group, on diminishing cancer-related fatigue in colorectal cancer survivors.

DETAILED DESCRIPTION:
The SoFiT study is a randomized controlled trial examining the effects of a behaviour change guided lifestyle intervention on increasing adherence to the World Cancer Research Fund (WCRF) cancer prevention guidelines, compared to the wait-list usual care group, on diminishing cancer-related fatigue in colorectal cancer survivors.

Colorectal cancer survivors who completed treatment six months to five years ago and who suffer from cancer-related fatigue, are randomized into two parallel groups: an intervention group or the wait-list usual care group. The intervention group follows a six-month personalized lifestyle program, which is guided by behaviour change techniques, to increase adherence to the World Cancer Research Fund cancer prevention guidelines on healthy nutrition, physical activity and healthy weight. Participants are guided by a lifestyle coach specialized in behaviour change. The wait-list usual care group receives a lifestyle program after the intervention period of six months: this includes two personalized behavioural coaching sessions and any material that the intervention group also received.

Both groups participate in measurements at baseline, three months, at the end of the intervention (six months) and at follow-up (twelve months). The follow-up timepoint is included to study long-term behavioural lifestyle change. The primary outcome is the change in cancer-related fatigue, as measured by the FACIT-Fatigue questionnaire, between the intervention and wait-list usual care group from baseline till six months.

Secondary outcomes include cancer-related fatigue (at other timepoints), skeletal muscle fat infiltration and cross-sectional area, gut microbiota composition, health-related quality of life, physical performance, sleep quality and duration, depression and anxiety, behavioural determinants and adherence to the WCRF guidelines by assessing habitual dietary intake, physical activity level, height, weight, waist circumference and BMI. Other outcomes of interest include, blood pressure, chrono-nutrition, colorectal cancer related complaints, hemoglobin blood levels, self-reported weight (at three months) and cost-effectiveness evaluation. Moreover, the following data will be collected to characterize the population: sociodemographic information (age, sex, marital status, education, smoking) and clinical parameters (time since diagnosis, current and received treatment, comorbidities, medicine and supplement use).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above.
* Completed curative stage I-III colorectal cancer treatment in the previous 6 months to 5 years.
* Live on a reasonable distance from the research center at the Wageningen University & Research (WUR) (i.e. maximum of ± 1 hour away).
* Classified as suffering from CRF through the Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale questionnaire with cut-off score below 34 indicating fatigue.
* Willingness to be randomized into either the intervention or wait-list control group.
* Willing and able to follow the lifestyle intervention.
* Able to understand and provide informed consent in Dutch.

Exclusion Criteria:

* Planning to participate or participating in another medical research that could possibly interfere with the study results.
* Excessive alcohol consumption (i.e. more than 4 glasses per day).
* Chronic drug use and unwillingly to stop using drugs.
* Unable/unwilling to comply with the intervention (e.g. through dementia, Alzheimer or mental illness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in cancer-related fatigue | Baseline till six months
  Cancer-related fatigue is assessed with the FACIT-Fatigue Scale, a 13 item questionnaire with scores ranging from 0-52. A score below 34 indicates fatigue. The minimal clinically important difference is reported to be 3.0 for this scale.

SECONDARY OUTCOMES:
Cancer-related fatigue | Twelve months
  Cancer-related fatigue is assessed with the FACIT-Fatigue Scale, a 13 item questionnaire with scores ranging from 0-52. A score below 34 indicates fatigue. The minimal clinically important difference is reported to be 3.0 for this scale.
Skeletal muscle fat infiltration and muscle circumference | Baseline and six months
  Echo intensity of the skeletal muscle rectus femoris, lateral gastrocnemius and biceps brachialis is measured using a portable ultrasound machine.
Gut microbiota composition | Baseline and six months
  Faecal samples are collected and the microbiota composition in this will be analyzed. The investigators will use 16S rRNA sequencing data for the taxonomic characterization of the gut microbiota. Eventually shotgun sequencing may also be done.
Health-related quality of life | Baseline and six months
  Health-related quality of life is measured with the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire, which contains the following domains of well-being: physical, social/family, emotional and functional. The 27-item questionnaire has scores ranging from 0 to 108.
Physical performance (3-minute step test) | Baseline and six months
  This test indicates cardiovascular fitness by heart rate measurement for one minute after the completion of three minutes of stepping.
Physical performance (5 times sit-to-stand test) | Baseline and six months
  This test indicates lower extremity skeletal muscle strength. The time necessary to achieve the standing position on the 5th repetition is measured.
Physical performance (tandem test) | Baseline and six months
  This test measures balance for three different standing positions. Each position has to be maintained for 10 seconds in order to pass the test.
Physical performance (chair sit-and-reach test) | Baseline and six months
  This test measures lower extremity and lower back flexibility. Participants sit on a chair and bend forward and reach for their toes. The distance between the hand and toes is measured.
Physical performance (strength: hand dynamometer) | Baseline and six months
  This test uses a hand dynamometer to measure strength.
Sleep quality and duration (Pittsburgh Sleep Quality Index) | Baseline, six months and 12 months
  Sleep quality is measured with the Pittsburgh Sleep Quality Index (PSQI), a 19-item questionnaire with scores ranging from 0-21. A score above 5 indicates bad sleep quality.
Sleep quality and duration (Consensus sleep diary morning) | Baseline and six months
  The Consensus sleep diary morning (CSD), a 15-item diary, is used for measuring other sleep outcomes such as sleep onset latency and sleep duration.
Depression | Baseline and six months
  Depression is measured using the 8-item Patient Healthcare Questionnaire (PHQ-8). It contains 8 items, and scores range from 0-24, with higher scores indicating a higher chance of depression.
Anxiety | Baseline and six months
  Anxiety is measured using the 7-item Generalized Anxiety Disorder (GAD-7). The GAD-7 contains 7 items, its scores range from 0-21, with higher scores indicating a higher chance of anxiety.
Behavioural determinants | Baseline, three months, six months and twelve months.
  Identified behavioural determinants through focus groups and a systematic review, are assessed using a self-reported questionnaire with questions based on previous reported questions on different determinants. These were adapted to reflect the WCRF guidelines. Higher scores for each of the determinants (scale 1-7) indicate better results.
Habitual dietary intake (Food Frequency Questionnaire) | Baseline, six months and twelve months
  Nutritional intake is measured using a semi-quantitative Food Frequency Questionnaire (FFQ). Scores are calculated using the Dutch National Food Consumption tables. In addition, the validated questionnaire Eetscore is used, which contains a short online questionnaire (10-15 minutes) that serves as an indicator to assess diet quality, based on the Dutch Healthy Diet index 2015 (DHD15-index). Scores range from 0-160, with higher scores indicating better diet quality.
Habitual dietary intake (Eetscore) | Baseline, three months, six months and twelve months
  Nutritional intake is also measured using the validated questionnaire Eetscore, which uses a short online questionnaire (10-15 minutes) that serves as an indicator to assess diet quality, based on the Dutch Healthy Diet index 2015 (DHD15-index). Scores range from 0-160, with higher scores indicating better diet quality.
Physical activity level (Short QUestionnaire to ASsess Health-enhancing physical activity) | Baseline, three months, six months and twelve months
  Physical activity is measured using the Short QUestionnaire to ASsess Health-enhancing physical activity (SQUASH). The questions in the SQUASH are pre-structured in commuting, leisure time, household and work/school activities. Scores will be assigned to the different reported activities base on intensities in MET and translated to minutes of physical activity.
Physical activity level (Accelerometer) | Baseline and six months
  Physical activity is also measured using ActivPalTM Micro3, an accelerometer measuring sedentary behaviour and physical activity. The ActivPalTM is worn for 9 days.
Anthropometric measurements (Height) | Baseline and six months
  Height (in cm) is measured with a stadiometer.
Anthropometric measurements (Weight) | Baseline, three months (self-reported) and six months
  Weight (in kg) is measured with a calibrated scale.
Anthropometric measurements (Waist circumference) | Baseline and six months
  Waist circumference (in cm) is measured using tape measures.
Cost-effectiveness evaluation | Baseline, three months and six months
  The cost-effectiveness of the intervention is evaluated using a questionnaire that includes items on for example costs that the participant has made in order to follow the lifestyle program.

OTHER OUTCOMES:
Blood pressure | Baseline and six months
  Blood pressure is measured using a sphygmomanometer. Both diastolic and systolic blood pressure are measured.
Heart rate | Baseline and six months
  Heart rate is measured using a sphygmomanometer.
Chrono-nutrition | Baseline and six months
  Chrono-nutrition, the timing of dietary intake, is measured with the "Chromes vragenlijst patiënten eetpatronen". This is a Dutch questionnaire containing 26 items that assess meal regularity (8-items), meal frequency (7-items), and meal clock time (11-items).
Colorectal cancer related complaints | Baseline and six months
  Measuring colorectal cancer specific problems is done using the additional concerns (i.e. subscale) of the Functional Assessment of Cancer Therapy - Colorectal (FACT-C). This questionnaire contains 9 items and scores are ranging from 0-28 points.
Hemoglobin levels | Baseline and six months
  Finger prick blood sampling is used for assessing haemoglobin status as an indicator for anaemia.
Sociodemographic information | Baseline (and six months)
  Sociodemographic information is collected using standardized questionnaires.
Clinical parameters | Baseline (and six months)
  Clinical parameters such as time since diagnosis, current and received treatment, comorbidities and medicine use, are collected either via standardized questionnaires or from medical records (part of informed consent).

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vries-Ten Have J, Manusama K, Verkaar AJCF, Beijer S, Sommeijer DW, Kampman E, Winkens LHH, Winkels RM. A randomised controlled intervention trial to study the effect of a personalised lifestyle programme on cancer-related fatigue among colorectal cancer survivors: protocol for the SoFiT study. Br J Nutr. 2024 Jul 28;132(2):248-258. doi: 10.1017/S0007114524001107. Epub 2024 May 28. PMID 38804183